CLINICAL TRIAL: NCT01234025
Title: A Phase 1b/2 Study of Docetaxel and Prednisone, With or Without ISIS 183750 (an eIF4E Inhibitor), in Patients With Castrate-Resistant Prostate Cancer
Brief Title: Safety and Tolerability Study of ISIS EIF4E Rx in Combination With Docetaxel and Prednisone (CRPC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 183750-CS3
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Castrate-Resistant Prostate Cancer
Keywords: Castrate-Resistant Prostate Cancer
MeSH Terms: interventions — Prednisone; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- Part 1 Cohort 1 (Experimental)
  Interventions: Drug: ISIS EIF4E Rx; Drug: Prednisone; Drug: Docetaxel
- Part 1 Cohort 2 (Experimental)
  Interventions: Drug: ISIS EIF4E Rx; Drug: Prednisone; Drug: Docetaxel
- Part 2 Arm A (Experimental)
  Interventions: Drug: Prednisone; Drug: Docetaxel
- Part 2 Arm B (Experimental)
  Interventions: Drug: ISIS EIF4E Rx; Drug: Prednisone; Drug: Docetaxel

INTERVENTIONS:
Drug: ISIS EIF4E Rx — 800 mg ISIS EIF4E Rx administered as a 3-hour intravenous infusion on Days 1, 8 and 15 of each 21 day cycle.
  Arms: Part 1 Cohort 1
Drug: ISIS EIF4E Rx — 1000 mg ISIS EIF4E Rx administered as a 3-hour intravenous infusion on Days 1, 8 and 15 of each 21 day cycle.
  Arms: Part 1 Cohort 2
Drug: ISIS EIF4E Rx — (Dose identified in Part 1)ISIS EIF4E Rx administered as a 3-hour intravenous infusion on Days 1, 8 and 15 of each 21 day cycle.
  Arms: Part 2 Arm B
Drug: Prednisone — 5 mg administered orally twice daily on days 1, 8, 15 and 22 of each cycle
Drug: Docetaxel — 75 mg/m2 administered as a 1-hour intravenous infusion on day 1 of each cycle

SUMMARY:
The purpose of this study is to examine the safety, tolerability and progression-free survival of patients with Castrate-Resistant Prostate Cancer treated with ISIS EIF4E Rx in combination with docetaxel and prednisone.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to Screening.
* Age ≥ 18 years.
* Histological or cytological diagnosis of adenocarcinoma of the prostate.
* Metastatic disease for which no curative therapy exists and for which systemic chemotherapy is indicated.
* Progression of disease despite either medical or surgical castration. If the patient received medical androgen ablation, a castrate level of testosterone (> or = 50 ng/dL) must have been present concurrent with disease progression. Progressive disease is defined as any one of the following:

  * Rising serum PSA levels: two consecutive increases in PSA levels documented over a previous reference value obtained at least one week apart with the value of the third point being ≥ 2 ng/mL. If the third PSA level is less than the second, an additional fourth test to confirm a rising PSA (i.e., the fourth value is ≥ the second value and is ≥ 2 ng/mL) is acceptable.
  * Progressive measurable disease defined as an increase in the sum of the diameters of measurable lesions over the smallest sum observed or the appearance of one or more new lesions as assessed by CT scan.
  * Bone progressions: appearance of 2 or more new lesions on bone scan or other imaging.
* If patient did not have a surgical orchiectomy:

  * The patient must be on androgen suppression treatment (e.g. LHRH agonist), have a castrate level of testosterone (< or = 50 ng/dL), and must be willing to continue the treatment throughout the study.
  * The patient must have discontinued treatment with anti-androgens (discontinued ≥ 4 weeks for flutamide and ≥ 6 weeks for nilutamide or bicalutamide prior to Screening) and have documented disease progression following discontinuation.
* PSA > or = 2 ng/mL during the Screening period.
* Performance status of 0 or 1 on the ECOG Performance Status Scale.
* Have an estimated life expectancy of at least 12 weeks.
* Adequate organ function within 14 days prior to first study dose (ISIS EIF4E Rx or docetaxel, whichever occurs first) including the following:

  * Absolute neutrophil count (ANC) > or = 1.5 x 109/L.
  * Platelet count > or = 100 x 109/L.
  * Total bilirubin < or = 1.0 x upper limit of normal (ULN).
  * Aspartate aminotransferase (AST) < or = 1.5 x ULN.
  * Alanine aminotransferase (ALT) < or = 1.5 x ULN.
  * Serum creatinine < or = 1.5 x ULN.
  * Prothrombin time (PT) and international normalized ratio (INR) within normal limits.
  * Activated partial thromboplastin time (aPTT) within normal limits.
* Part 1: Have had no more than 1 prior chemotherapy or biological therapy regimen (approved or experimental; all previous hormonal therapies are allowed and not counted as biological therapy for this inclusion criterion) for prostate cancer. This does not include treatments that may have been received in the adjuvant or neoadjuvant setting. A regimen is defined as two or more consecutive cycles of treatment. Part 2: Have had no prior chemotherapy or biological therapy (approved or experimental; all previous hormonal therapies are allowed and not counted as biological therapy for this inclusion criterion) in any setting for prostate cancer.
* Have discontinued all previous therapies for cancer (except treatment with LHRH analogues) as follows:

  * Part 1: cytotoxic chemotherapy must be discontinued at least 4 weeks prior to screening; Part 2: see Inclusion Criteria 11.
  * Part 1: biological treatment (other than hormonal treatments) must be discontinued for at least 6 weeks prior to screening; Part 2: see Inclusion Criteria 11.
  * Hormone therapies (e.g., abiraterone, MDV3100) must have been discontinued 4 weeks prior to screening.
  * Radiotherapy must be discontinued at least 4 weeks prior to screening, and the patient must have recovered from the acute effects of therapy.
* Recovery from all toxicities of prior therapy to ≤ Grade 2 by NCI CTCAE, version 4.0 (Exception: any toxicity that in the view of the Investigator is not a clinically significant safety risk for further therapy administration, including, but not limited to: anemia, fatigue, erectile dysfunction, hot flashes, lymphedema of an extremity, dizziness, cough, and urinary incontinence).
* Men of reproductive potential must agree to use an effective form of contraception, as determined by the Investigator, during the treatment period of the study and for 10 weeks following the last dose of study drug.
* The patient is willing and able to comply with the study visit schedule and procedures, and geographic proximity (Investigator's discretion) that allows adequate follow-up.

Exclusion Criteria:

* Treatment with another investigational drug or device within 4 weeks or biological agent within 6 weeks before Screening or 5 half-lives of study agent, whichever is longer.
* Pre-existing peripheral neuropathy > or = Common Terminology Criteria for Adverse Events, Version 4.0 (CTCAE) Grade 2.
* Patients with treated or untreated parenchymal brain metastases or leptomeningeal disease. Currently active malignant epidural disease is also excluded. Previously treated epidural disease does not exclude the patient from the study. (Note: CT or MRI of brain is not needed to rule these out unless the patient has clinical symptoms suggestive of CNS metastases).
* Have active infection or serious concomitant systemic disorder (for example, heart failure) incompatible with the study (at the discretion of the Investigator).
* Presence or history of other malignancies except non-melanoma skin cancer or solid tumors curatively treated at least 5 years previously with no subsequent evidence of recurrence.
* Presence of an underlying disease state associated with active bleeding.
* Ongoing therapy with oral or parenteral anticoagulants (e.g., heparin, warfarin/coumadin). Low-dose anticoagulants for maintenance of catheter patency and low dose aspirin (≤ 325 mg/day) and nonsteroidal antiinflammatory agents are not exclusionary.
* Concurrent treatment with other anticancer drugs.
* Inability to comply with protocol or study procedures.
* Previous therapy with strontium or samarium.
* Patients who have had irradiation of ≥ 25% of the bone marrow (e.g. pelvic irradiation).
* Use of any herbal products, including saw palmetto within 1 week of screening and throughout the study.
* Initiation of treatment with bisphosphonates, or change in dose, within 4 weeks of assignment to dosing in this study. Patients taking bisphosphonates should not have their dosing regimen altered during the study unless medically warranted.
* Known history of HIV, HCV, or chronic HBV infection.
* Previous treatment with a therapeutic antisense oligonucleotide or siRNA.
* Planned concomitant participation in another clinical trial of an experimental agent, vaccine, or device.
* Have any other medical conditions that, in the opinion of the Investigator, would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2010-11; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | At the end of each 21 day cycle

CONTACTS AND LOCATIONS:
Locations (38):
- United States (11):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - San Bernardino Urological Associates, San Bernardino, California
  - Fort Range Cancer Center, Fort Collins, Colorado
  - Norwalk Hospital- Whittingham Cancer Center, Norwalk, Connecticut
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - University of Miami, Miller School of Medicine - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Central Baptist Hospital Clinical Research Center, Lexington, Kentucky
  - Feist-Weiller Cancer Center, Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - St. Luke's - Roosevelt Hospital Center, New York, New York
  - James P. Wilmont Cancer Center - University of Rochester Medical Center, Rochester, New York
  - Gabrail Cancer Center, Canton, Ohio
- Hungary (5):
  - Szent Janos Hospital and Unified Hospitals of North Buda, Budapest
  - Semmelweis University Faculty of Medicine, Budapest
  - National Institute of Oncology, Budapest
  - University of Pecs, Institute of Oncology, Pécs
  - Fejer County St. Gyorgy Hospital, Dept of Oncology, Székesfehérvár
- Poland (6):
  - Ewa Pilecka Clinical Oncology Department and Outpatient Chemotherapy Unit, Bialostockie M.Sklodowska-Curie Oncology Centre in Bialystok, Bialystok
  - Regionalny Szpital Specjalistyczny im. dr Wladyslawa Bieganskiego, Oddzial Onkologii Klinicznej, Grudziądz
  - Department of Chemotherapy, Health Care Facility of the Ministry of Internal Affairs and Administration and Warminsko-Mazurskie Oncology Centre in Olsztyn, Olsztyn
  - Clinical Oncology Department and Day Hospitalization Unit, Independent Public Healthcare Facility T. Koszarowski Opolskie Oncology Centre in Opole, Opole
  - Department of Urologic Oncology, Maria Sklodowska-Curie Institute of Oncology, Warsaw
  - Clinical Oncology Department/Chemotherapy Department, MAGODENT Non-Public Healthcare Facility, Branch Facility No. 4, Warsaw
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico
- Romania (8):
  - Alba Lulia Emergency County Hospital, Alba Iulia
  - Dr Constantin Opris Emergency County Hospital, Baia Mare
  - S.C. Rapid Diagnosis Polyclinic SRL, Brasov
  - Fundeni Clinical Institute, Bucharest
  - "Prof. Dr Th Burghele" Clinical Hospital, Bucharest
  - SC Medisprof SRL, Cluj-Napoca
  - S.C. Provita 2000 SRL, Constanța
  - SC Oncolab SRL, Medical Oncology Dept, Craiova
- Russia (7):
  - State Therapeutical and Prophylactic Institution: Chelyabinsk Regional Clinical Oncology Center, Chemotherapy Department, Chelyabinsk
  - State Medical Institution: Kursk Regional Oncological Center, Chemotherapy Dept, Kursk
  - State Medical Institution of the City of Moscow: Municipal Clinical Hospital #57 under Moscow Department for Healthcare, Moscow
  - Non-State Medical Institution: Central Clinical Hospital #2 n.a. N.A. Semashko under OJSC Russian Railways, Chemotherapy Dpmt, Moscow
  - Federal State Budget Institution: "Medical Radiological Research Center" under the Ministry of Health Care and Social Development of the Russian Federation, Obninsk
  - St. Petersburg State Medical Institution: St. Petersburg Municipal Oncological Center, Department of Urologic Oncology, Saint Petersburg
  - Russian Research Center for Radiology and Surgical Technologies, Saint Petersburg